CLINICAL TRIAL: NCT06639828
Title: A Phase 4, Open-Label, Non-randomised, Multicentre Study to Evaluate Safety and Efficacy of Intravenous Administration of Sonazoid™ for Contrast-Enhanced Ultrasound Liver Imaging in Paediatric Patients
Brief Title: Phase 4 Paediatric Study to Evaluate Sonazoid Safety and Efficacy for Contrast-Enhanced Ultrasound Liver Imaging
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: PPD Development, LP (Industry); Medidata Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-045-401; 1007450 (Other: IRAS ID); 2023-505569-95-00 (Other: EU CT)
Record Dates: First submitted 2024-10-01; First posted 2024-10-15 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Focal Liver Lesions
Keywords: Contrast-Enhanced Ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sonazoid (Experimental): Participants will receive a single iv dose of Sonazoid™, dosed according to body weight (0.12 μL microbubbles/kg)
  Interventions: Diagnostic Test: Contrast-Enhanced Ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast-Enhanced Ultrasound — Following unenhanced (pre-contrast) ultrasound imaging of the target focal liver lesions (FLL), Sonazoid™ will be intravenously administered and a contrast-enhanced examination will be performed.

SUMMARY:
Liver tumours, 40% of which are benign, account for 1% to 4% of all solid tumours in children. The benign tumours are mainly haemangiomas, liver hamartomas, and liver cell adenomas. The malignant tumours are mainly hepatoblastoma, hepatocellular carcinoma (HCC), malignant liver mesothelioma, and rhabdomyosarcoma. The differential diagnosis of liver masses in children is generally based on the child's age, the clinical evaluation (including alpha-fetoprotein test results), and imaging characteristics.

Liver tumours seldom produce clear symptoms and signs in the early stages, and they progress rapidly. As a result, most liver tumours are not diagnosed until the middle or late stages. To improve survival among patients with liver tumours, clinicians must find the liver tumours as early as possible and determine whether the tumours are benign or malignant. Conventional ultrasonography is commonly used for screening, and is preferred as the first-line imaging technique for children. Not only does it have a wide range of applications and a high diagnostic yield, but it is well accepted by patients and their parents. It can be performed in the examination room with the parents present, allowing real-time imaging and direct interaction with patient and parents.

CEUS is a non-invasive imaging technology that can continuously and dynamically observe blood perfusion in tumours in real-time through injection of a contrast agent to enhance the blood flow reflux signal in the human body. Consequently, CEUS is useful for visualising capillaries and tissue perfusion in the human body.

The purpose of this current study is to evaluate the use of Sonazoid™ perfluorobutane (PFB) microbubbles as a contrast medium for CEUS for evaluation of solitary liver masses in children.

DETAILED DESCRIPTION:
This Phase 4, open-label, non-randomised, multicentre prospective study in Europe will enrol paediatric patients who are presenting with ≥1 confirmed untreated target FLL. This study plans to enrol at least 50 subjects at up to 12 centres in Europe. If a patient has multiple FLLs, the Investigator must select the target lesion at their discretion. Where possible, the target lesion should be a clearly visible and accessible lesion that could be easily followed during the non-CE ultrasound examination and all phases of the CEUS examination. The reference diagnosis/standard of truth for the target lesion of interest will be established by the principal investigators/sub-investigators on the basis of all available clinical information, including the results of biopsy, if available, and the dynamic CECT or CEMRI examination required for the study.

Following unenhanced (pre-contrast) ultrasound imaging of the target FLL, a single dose of Sonazoid™, dosed according to body weight (0.12 μL microbubbles/kg), will be intravenously administered to each patient, and a CEUS examination will be performed, with images acquired as specified in the Imaging Manual.

The unenhanced ultrasound and CEUS images will be assessed by 3 independent blinded readers following WFUMB-EFSUMB guidelines for adults, and in accordance with the Independent Review Charter. The diagnoses based on the unenhanced ultrasound and the CEUS results will be compared with the reference diagnosis/standard of truth for the target lesion. The diagnostic accuracy, sensitivity and specificity of the unenhanced ultrasound and CEUS images will then be calculated. Clinical safety data will be collected throughout the study. Safety will be evaluated by monitoring subjects for the occurrence of AEs.

ELIGIBILITY:
Inclusion Criteria:

* The subject is <18 years of age on the day of consent.
* The subject has at least 1 untreated FLL with ≤8 lesions (excluding cysts), with ≤8 cm confirmed in a diagnostic examination performed in the past month (or past 3 months if the lesion was benign) and that could also be visualised when obtained via unenhanced ultrasound imaging
* The subject has had a dynamic CECT or CEMRI examination within the past month or is scheduled to have one in the month following inclusion in the study, and these images are/would be available.
* The subject can comply with study procedures.
* Parents or legally authorised representatives have signed the Informed Consent Form approved for this study by the Independent Review Board (IRB)/Independent Ethics Committee (IEC). The form will indicate that the patient (and/or a legally acceptable representative) has been informed of all pertinent aspects of the study. Patients who are able to provide assent have signed an age-appropriate paediatric assent form
* Post-menarcheal female patients must have a negative urine pregnancy test at screening and at pre-dose on the dosing day.
* Post-menarcheal female patients and male patients who are sexually active with a partner of childbearing potential must be practicing abstinence or be using an effective form of birth control (See Section 8.6) for ≥30 days before being enrolled in the study
* The subject has a body weight of 3 kg or greater.
* The subject has a negative egg allergy test if the egg allergy status of the subject is unknown.

Exclusion Criteria:

* The subject has a known or suspected hypersensitivity to any of the components of Sonazoid™, including a history of allergies to eggs or egg products (i.e., manifested by full body rash, respiratory difficulty, oral or laryngeal swelling, hypotension, or shock).
* The subject has an acute clinically fatal condition (i.e., the expected survival is ≤6 months).
* The subject has previously received Sonazoid™ or another ultrasound contrast agent within the past 30 days.
* The subject had undergone or is planning to undergo an examination with a contrast agent (i.e., iodinated x-ray contrast agent, MRI contrast agent or another ultrasound contrast agent) within the 24 hours before or after Sonazoid™ injection.
* The subject has undergone or was undergoing systemic or loco-regional chemotherapy or radiation therapy
* The subject is participating in another clinical trial with an unregistered medicinal product, or less than 30 days has passed since the subject completed participation in such a trial
* The subject is a pregnant or lactating female.
* The physician judges that a large-enough needle (24-gauge or larger) cannot be inserted.
* The subject has a known right-left cardiac shunt.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Sonazoid-enhanced ultrasound at imaging focal liver lesions during the vascular phase of imaging | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 4-minutes post injection for the vascular phase] and blinded image evaluations shall be executed remotely at a central lab
  Accuracy of the diagnosis based on the independent blinded read of the Sonazoid™-enhanced imaging for lesion differentiation (benign or malignant FLLs) during vascular phase imaging. The WFUMB-EFSUMB guidelines for interpreting CEUS of the liver in adults shall be used for interpreting the images and the subject's baseline diagnosis (well-established by CECT, CEMRI or biopsy) will be used as the reference diagnosis/standard of truth.
Sensitivity of Sonazoid-enhanced ultrasound at imaging focal liver lesions during the vascular phase of imaging | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 4-minutes post injection for the vascular phase] and blinded image evaluations shall be executed remotely at a central lab
  Sensitivity of the diagnosis based on the independent blinded read of the Sonazoid™-enhanced imaging for lesion differentiation (benign or malignant FLLs) during vascular phase imaging. The WFUMB-EFSUMB guidelines for interpreting CEUS of the liver in adults shall be used for interpreting the images and the subject's baseline diagnosis (well-established by CECT, CEMRI or biopsy) will be used as the reference diagnosis/standard of truth.
Specificity of Sonazoid-enhanced ultrasound at imaging focal liver lesions during the vascular phase of imaging | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 4-minutes post injection for the vascular phase] and blinded image evaluations shall be executed remotely at a central lab
  Specificity of the diagnosis based on the independent blinded read of the Sonazoid™-enhanced imaging for lesion differentiation (benign or malignant FLLs) during vascular phase imaging. The WFUMB-EFSUMB guidelines for interpreting CEUS of the liver in adults shall be used for interpreting the images and the subject's baseline diagnosis (well-established by CECT, CEMRI or biopsy) will be used as the reference diagnosis/standard of truth.

SECONDARY OUTCOMES:
Comparison of accuracy of Sonazoid-enhanced ultrasound to Unenhanced ultrasound at imaging focal liver lesions during vascular phase | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 4-minutes post injection for the vascular phase] and blinded image evaluations shall be executed remotely at a central lab.
  Accuracy of the diagnosis (benign or malignant FLL) based on the Sonazoid™-enhanced imaging by vascular phase imaging, as compared with the unenhanced ultrasound imaging, when the baseline diagnosis is used as the reference standard.
Comparison of accuracy of Sonazoid-enhanced ultrasound to Unenhanced ultrasound at imaging focal liver lesions during vascular and Kupffer phase | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 10-minutes post injection for the vascular and Kupffer phase(s)] and blinded image evaluations shall be executed remotely at a central lab
  Accuracy of the diagnosis (benign or malignant FLL) based on the Sonazoid™-enhanced imaging by vascular phase and Kupffer phase imaging, as compared with the unenhanced ultrasound imaging, when the baseline diagnosis is used as the reference standard.
Comparison of sensitivity of Sonazoid-enhanced ultrasound to Unenhanced ultrasound at imaging focal liver lesions during vascular phase | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 4-minutes post injection for the vascular phase] and blinded image evaluations shall be executed remotely at a central lab.
  Sensitivity of the diagnosis (benign or malignant FLL) based on the Sonazoid™-enhanced imaging by vascular phase imaging, as compared with the unenhanced ultrasound imaging, when the baseline diagnosis is used as the reference standard.
Comparison of sensitivity of Sonazoid-enhanced ultrasound to Unenhanced ultrasound at imaging focal liver lesions during vascular and Kupffer phase | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 10-minutes post injection for the vascular and Kupffer phase(s)] and blinded image evaluations shall be executed remotely at a central lab
  Sensitivity of the diagnosis (benign or malignant FLL) based on the Sonazoid™-enhanced imaging by vascular phase and Kupffer phase imaging, as compared with the unenhanced ultrasound imaging, when the baseline diagnosis is used as the reference standard.
Comparison of specificity of Sonazoid-enhanced ultrasound to Unenhanced ultrasound at imaging focal liver lesions during vascular phase | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 4-minutes post injection for the vascular phase] and blinded image evaluations shall be executed remotely at a central lab.
  Specificity of the diagnosis (benign or malignant FLL) based on the Sonazoid™-enhanced imaging by vascular phase imaging, as compared with the unenhanced ultrasound imaging, when the baseline diagnosis is used as the reference standard.
Comparison of specificity of Sonazoid-enhanced ultrasound to Unenhanced ultrasound at imaging focal liver lesions during vascular and Kupffer phase | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 10-minutes post injection for the vascular and Kupffer phase(s)] and blinded image evaluations shall be executed remotely at a central lab
  Specificity of the diagnosis (benign or malignant FLL) based on the Sonazoid™-enhanced imaging by vascular phase and Kupffer phase imaging, as compared with the unenhanced ultrasound imaging, when the baseline diagnosis is used as the reference standard.
Comparison of diagnostic confidence of Sonazoid-enhanced ultrasound to Unenhanced ultrasound at imaging focal liver lesions during vascular phase | Images to be captured during the studies CEUS examination [approximately 5 seconds prior to bolus injection, up to 4-minutes post injection for the vascular phase] and blinded image evaluations shall be executed remotely at a central lab.
  The difference in the diagnostic confidence for the unenhanced ultrasound imaging and that for the Sonazoid™-enhanced ultrasound imaging based on the vascular phase. The difference in the diagnostic confidence will ranged from -3 to 3, higher scores mean better outcome.
Safety of Sonazoid following intravenous administration of IMP in paediatric patients based on Treatment-emergent adverse events | From administration of Sonazoid, up to 4 hours for in-person monitoring followed by 24-hour and 72-hour telephone follow ups
  Number and percentage of subjects with Treatment-emergent adverse events, defined as adverse events that occurred at any timepoint from the administration of Sonazoid™ to the end of the study (72 hours after Sonazoid™ administration)
Safety of Sonazoid following intravenous administration of IMP in paediatric patients based on drug-related Treatment-emergent adverse events | From administration of Sonazoid, up to 4 hours for in-person monitoring followed by 24-hour and 72-hour telephone follow ups
  Number and percentage of subjects with drug-related Treatment-emergent adverse events
Safety of Sonazoid following intravenous administration of IMP in paediatric patients based on Treatment-emergent Serious Adverse events | From administration of Sonazoid, up to 4 hours for in-person monitoring followed by 24-hour and 72-hour telephone follow ups
  Number and percentage of subjects with Treatment-emergent Serious Adverse events
Safety of Sonazoid following intravenous administration of IMP in paediatric patients based on Physical examination | Pre-administration of Sonazoid and 4 hours post administration
  Number and percentage of subjects with changes in physical examination status (normal/abnormal)
Safety of Sonazoid following intravenous administration of IMP in paediatric patients based on Vital signs | Pre-administration of Sonazoid and 4 hours post administration
  Summary statistics of systolic/diastolic blood pressure, heart rate, respiratory rate, body temperature, and oxygen saturation for each timepoint
Safety of Sonazoid following intravenous administration of IMP in paediatric patients based on Clinical laboratory results | Pre-administration of Sonazoid and 4 hours post administration
  Summary statistics of clinical laboratory for each timepoint

CONTACTS AND LOCATIONS:
Overall Officials: David Thompson, Study Director — GE Healthcare
Locations (6):
- Munich University Hospital, München, Germany
- Italy (2):
  - Papa Giovanni XXIII Hospital, Bergamo
  - Giannina Gaslini Institute, Genoa
- United Kingdom (3):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - King's College Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No